CLINICAL TRIAL: NCT04210843
Title: A Multi-center, Double-blinded and Open-label Extension Study to Evaluate the Efficacy and Safety of Ligelizumab as Retreatment, Self-administered Therapy and Monotherapy in Chronic Spontaneous Urticaria Patients Who Completed Studies CQGE031C2302, CQGE031C2303, CQGE031C2202 or CQGE031C1301
Brief Title: Study of Efficacy and Safety of Ligelizumab in Chronic Spontaneous Urticaria Patients Who Completed a Previous Study With Ligelizumab
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was terminated due to a strategic decision by Novartis to discontinue development of ligelizumab in CSU. This decision was not based on any safety concerns.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CQGE031C2302E1; 2019-001792-37 (EudraCT Number)
Record Dates: First submitted 2019-12-17; First posted 2019-12-26 (Actual); Results first posted 2023-07-13 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Chronic Spontaneous Urticaria
Keywords: Anti-IgE; chronic spontaneous urticaria; hives severity score; itch severity score; urticaria activity score; CSU
MeSH Terms: conditions — Chronic Urticaria | interventions — ligelizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants transitioning from CQGE031C2302 (NCT03580369) and CQGE031C2303 (NCT03580356) were treated in a double-blind manner for the first 12 weeks of treatment. Thereafter, they were treated in an open-label manner.
  No blinding was required for participants transitioning from CQGE031C1301 (NCT03907878) and CQGE031C2202 (NCT03437278)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ligelizumab 72 mg LIVI -ligelizumab 120 mg PFS (Experimental): Participants received 72 mg of ligelizumab liquid in vial (LIVI) subcutaneously every 4 weeks for the first 12 weeks. Thereafter, participants received 120 mg of ligelizumab pre-filled syringe (PFS) subcutaneously every 4 weeks for up to 92 additional weeks (continuous or interrupted if the participant entered the observation period 2).
  Interventions: Drug: Ligelizumab
- Ligelizumab 120 mg LIVI -ligelizumab 120 mg PFS (Experimental): Participants received 120 mg of ligelizumab liquid in vial (LIVI) subcutaneously every 4 weeks for the first 12 weeks. Thereafter, participants received 120 mg of ligelizumab pre-filled syringe (PFS) subcutaneously every 4 weeks for up to 92 additional weeks (continuous or interrupted if the participant entered the observation period 2).
  Interventions: Drug: Ligelizumab

INTERVENTIONS:
Drug: Ligelizumab — For the first 12 weeks of treatment: i) participants transitioning from CQGE031C2302 (NCT03580369) and CQGE031C2303 (NCT03580356) previously treated with ligelizumab 72 mg LIVI s.c. Q4W were treated with the same dose regimen in a double-blind manner; ii) all other participants transitioning from CQGE031C2302 (NCT03580369) and CQGE031C2303 (NCT03580356) were treated with ligelizumab 120 mg LIVI s.c. Q4W in a double-blind manner; iii) participants transitioning from CQGE031C1301 (NCT03907878) and CQGE031C2202 (NCT03437278) were treated with ligelizumab 120 mg LIVI s.c. Q4W in an open-label manner.
  Thereafter, all participants were switched to ligelizumab 120 mg s.c. PFS Q4W in an open-label manner and they were offered an opportunity to self-administer ligelizumab.
  The longest possible treatment was 104 weeks, however this treatment might not be continuous and might span over a period of 156 weeks due to the possibility of entering the intervening observation period.
  Other Names: QGE031

SUMMARY:
The purpose of this extension study was to establish efficacy and safety of ligelizumab. This was assessed in adult and adolescent chronic spontaneous urticaria (CSU) patients who had completed a preceding ligelizumab study and have relapsed, following treatment in these preceding studies, despite standard of care H1-antihistamine (H1-AH) treatment.

This study also fulfilled the Novartis commitment to provide post-trial access to patients who had completed studies: CQGE031C2302 (NCT03580369), CQGE031C2303 (NCT03580356), CQGE031C2202 (NCT03437278) or CQGE031C1301 (NCT03907878).

DETAILED DESCRIPTION:
This was a Phase IIIb multi-center, double-blinded and open-label extension study to evaluate efficacy and safety of ligelizumab retreatment with H1-AHs background therapy with an option for ligelizumab monotherapy (i.e., discontinuation of background H1-AH) in adult and adolescent CSU participants who had completed one of the preceding studies, in the setting of retreatment and self-administration.

Participants with weekly urticaria activity score (UAS7) < 16 during screening entered the first (investigational treatment-free) observation period (OBS1), with a duration up to 36 weeks.

Participants with UAS7 ≥ 16 during screening or OBS1 were assigned to 1 of the 2 treatment arms and entered the treatment period (first half treatment period, referred to as TRT1). The first half treatment period (TRT1) was 52 weeks (from Week 0 to Week 52). Participants remained on the same H1-AH background medication they were taking in the preceding studies. TRT1 was divided into:

* The first 12 weeks in TRT1:

  i. participants transitioning from CQGE031C2302 (NCT03580369) and CQGE031C2303 (NCT03580356) previously treated with ligelizumab 72 mg liquid in vial subcutaneously (s.c.) every 4 weeks (Q4W) were treated with the same dose regimen in a double-blind manner in this extension study; ii. all other participants transitioning from CQGE031C2302 (NCT03580369) and CQGE031C2303 (NCT03580356) were treated with ligelizumab 120 mg liquid in vial s.c., Q4W, in a double-blind manner in this extension study; iii. participants transitioning from CQGE031C1301 (NCT03907878) and CQGE031C2202 (NCT03437278) were treated with ligelizumab 120 mg liquid in vial s.c., Q4W in an open-label manner in this extension study.
* After the first 12 weeks in TRT1 (and up to Week 52), all participants were switched to ligelizumab 120 mg s.c. pre-filled syringe (PFS) Q4W in an open-label manner and they were offered an opportunity to self-administer ligelizumab outside the clinic.

The second half of the treatment period (TRT2) was 52 weeks (from Week 52 to Week 104). Participants with UAS7>6 and <16 or with UAS7 ≥ 16 for whom the benefit-risk was deemed as positive by the investigator at Week 52 of TRT1 were transitioned to the TRT2 (ligelizumab 120 mg s.c. Q4W PFS) unless a decision to stop treatment was made based on a risk-benefit assessment. They were not allowed to discontinue H1- AH background medication.

Participants with UAS7 ≤ 6 at Week 52 of TRT1 entered the second (investigational treatment-free) observation period (OBS2) for up to 52 weeks and remained on the same H1-AH background medication they were taking in the preceding studies. Participants with UAS7 ≤ 6 at Week 52 of TRT1 who entered the second observation period (OBS2) and relapsed (UAS7 ≥ 16) were transitioned to the TRT2 and were also offered the opportunity to discontinue their H1-AH background medication (i.e. ligelizumab 120 mg s.c. q4w PFS monotherapy) after 12 weeks in TRT2. Participants who entered the OBS2 and did not relapse (UAS7<16) exited the study at the end of the OBS2 period.

Finally, participants who were in TRT2 entered the post-treatment follow-up period after treatment discontinuation, with duration of 12 weeks (for participants who did not complete a continuous 104-week treatment) or 52 weeks (for participants who completed the full 104-week treatment period without interruption). Participants who decided to remain on H1-AH background medication continued to use H1-AH background medication. Participants who decided to go off H1- AH background medication continued to remain off.

ELIGIBILITY:
Key Inclusion Criteria:

* Written informed consent
* Subjects who successfully completed all of the treatment period and the follow-up period in any of the following studies: CQGE031C2302 (NCT03580369), CQGE031C2303 (NCT03580356), CQGE031C2202 (NCT03437278) or CQGE031C1301 (NCT03907878)
* Male and female, adult and adolescent subjects ≥12 years of age
* Willing and able to complete a daily symptom eDiary for the duration of the study and adhere to the study visit schedule

Key Exclusion Criteria:

* Use of investigational drugs, other than those in use in the preceding studies, at the time of enrollment
* Use of omalizumab within 16 weeks of Screening
* History of hypersensitivity to the study drug ligelizumab or its components, or to drugs of similar chemical classes
* New onset or signs and symptoms of any form of chronic urticarias other than CSU during the preceding studies CQGE031C2302 (NCT03580369), CQGE031C2303 (NCT03580356) or CQGE031C2202 (NCT03437278).
* Diseases with possible symptoms of urticaria or angioedema
* Subjects with evidence of helminthic parasitic infection
* Documented history of anaphylaxis
* Pregnant or nursing (lactating) women

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1033 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (244):
- United States (39):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Gilbert, Arizona
  - Novartis Investigative Site, Litchfield Park, Arizona
  - Novartis Investigative Site, Scottsdale, Arizona
  - Novartis Investigative Site, Little Rock, Arkansas
  - Novartis Investigative Site, Bakersfield, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Redwood City, California
  - Novartis Investigative Site, San Jose, California
  - Novartis Investigative Site, Colorado Springs, Colorado
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Greenacres City, Florida
  - Novartis Investigative Site, Sarasota, Florida
  - Novartis Investigative Site, Tallahassee, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Boise, Idaho
  - Novartis Investigative Site, Evansville, Indiana
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Overland Park, Kansas
  - Novartis Investigative Site, Bangor, Maine
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, White Marsh, Maryland
  - Novartis Investigative Site, Ypsilanti, Michigan
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Rochester, Minnesota
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Missoula, Montana
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Toledo, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Tulsa, Oklahoma
  - Novartis Investigative Site, Clackamas, Oregon
  - Novartis Investigative Site, Medford, Oregon
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, North Charleston, South Carolina
  - Novartis Investigative Site, El Paso, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Murray, Utah
  - Novartis Investigative Site, Bellingham, Washington
- Argentina (12):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Ciudad Autonoma de Bs As, Buenos Aires
  - Novartis Investigative Site, La Plata, Buenos Aires
  - Novartis Investigative Site, Mendoza, Mendoza Province
  - Novartis Investigative Site, Buenos Aires, Nueve De Julio
  - Novartis Investigative Site, Santa Fe, Rosario
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Bahía Blanca
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, CABA
  - Novartis Investigative Site, Capital Federal
  - Novartis Investigative Site, Salta
- Australia (3):
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, East Melbourne, Victoria
  - Novartis Investigative Site, Parkville, Victoria
- Novartis Investigative Site, Vienna, Austria
- Belgium (4):
  - Novartis Investigative Site, Jette, Brussels Capital
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Loverval
- Brazil (6):
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Alphaville Barueri, São Paulo
  - Novartis Investigative Site, Santo André, São Paulo
  - Novartis Investigative Site, São José do Rio Preto, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Bulgaria (3):
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Varna
- Canada (6):
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Kingston, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Waterloo, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
- Chile (3):
  - Novartis Investigative Site, Vitacura, Santiago Metropolitan
  - Novartis Investigative Site, Osorno
  - Novartis Investigative Site, Santiago
- Novartis Investigative Site, Medellín, Antioquia, Colombia
- Novartis Investigative Site, Zagreb, Croatia
- Czechia (4):
  - Novartis Investigative Site, Teplice, CZE
  - Novartis Investigative Site, Prague, Prague 1
  - Novartis Investigative Site, Olomouc
  - Novartis Investigative Site, Pilsen
- Novartis Investigative Site, Copenhagen NV, Denmark
- Novartis Investigative Site, Tallinn, Estonia
- France (5):
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Pierre-Bénite
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Toulouse
- Germany (24):
  - Novartis Investigative Site, Bad Bentheim
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Langenau
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, Memmingen
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Osnabrück
  - Novartis Investigative Site, Stade
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Tübingen
- Novartis Investigative Site, Athens, Greece
- Novartis Investigative Site, Guatemala City, Guatemala
- Hungary (4):
  - Novartis Investigative Site, Kecskemét, Bács-Kiskun county
  - Novartis Investigative Site, Szeged, Csongrád megye
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Pécs
- India (7):
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Belagavi, Karnataka
  - Novartis Investigative Site, Mangalore, Karnataka
  - Novartis Investigative Site, Nashik, Maharashtra
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, New Delhi
  - Novartis Investigative Site, Vijayawada
- Israel (5):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Kfar Saba
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Rehovot
- Italy (4):
  - Novartis Investigative Site, Cagliari, CA
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Siena, SI
- Japan (18):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Ichikawa, Chiba
  - Novartis Investigative Site, Chikushino-shi, Fukuoka
  - Novartis Investigative Site, Hiroshima, Hiroshima
  - Novartis Investigative Site, Obihiro, Hokkaido
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Nishinomiya, Hyōgo
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kamimashi-gun, Kumamoto
  - Novartis Investigative Site, Neyagawa, Osaka
  - Novartis Investigative Site, Sakai, Osaka
  - Novartis Investigative Site, Izumo, Shimane
  - Novartis Investigative Site, Itabashi-ku, Tokyo
  - Novartis Investigative Site, Machida, Tokyo
  - Novartis Investigative Site, Setagaya-ku, Tokyo
  - Novartis Investigative Site, Shinagawa Ku, Tokyo
  - Novartis Investigative Site, Fukuoka
- Lebanon (3):
  - Novartis Investigative Site, Beirut
  - Novartis Investigative Site, El Achrafiyé
  - Novartis Investigative Site, Saida
- Malaysia (3):
  - Novartis Investigative Site, Kuala Lumpur, Kuala Lumpur
  - Novartis Investigative Site, Ipoh, Perak
  - Novartis Investigative Site, George Town, Pulau Pinang
- Mexico (2):
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Villahermosa, Tabasco
- Netherlands (3):
  - Novartis Investigative Site, Bergen op Zoom
  - Novartis Investigative Site, Breda
  - Novartis Investigative Site, Utrecht
- Novartis Investigative Site, Muscat, Oman
- Peru (2):
  - Novartis Investigative Site, Miraflores, Lima region
  - Novartis Investigative Site, San Borja, Lima region
- Philippines (2):
  - Novartis Investigative Site, City of Taguig, National Capital Region
  - Novartis Investigative Site, Pasig
- Poland (7):
  - Novartis Investigative Site, Ksawerów, POL
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Rzeszów
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Novartis Investigative Site, San Juan, Puerto Rico
- Romania (3):
  - Novartis Investigative Site, Bucharest, District 2
  - Novartis Investigative Site, Brasov
  - Novartis Investigative Site, Cluj-Napoca
- Russia (9):
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Rostov-on-Don
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Saratov
  - Novartis Investigative Site, Smolensk
  - Novartis Investigative Site, Stavropol
- Novartis Investigative Site, Singapore, Singapore
- Slovakia (8):
  - Novartis Investigative Site, Kežmarok
  - Novartis Investigative Site, Komárno
  - Novartis Investigative Site, Levice
  - Novartis Investigative Site, Nové Zámky
  - Novartis Investigative Site, Považská Bystrica
  - Novartis Investigative Site, Svidník
  - Novartis Investigative Site, Topoľčany
  - Novartis Investigative Site, Žilina
- South Africa (3):
  - Novartis Investigative Site, Cape Town, Western Province
  - Novartis Investigative Site, Cape Town
  - Novartis Investigative Site, Durban
- South Korea (8):
  - Novartis Investigative Site, Daegu, Dalseo Gu
  - Novartis Investigative Site, Wŏnju, Gangwon-do
  - Novartis Investigative Site, Hwaseong-si, Gyeonggi-do
  - Novartis Investigative Site, Suwon, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul, Seocho Gu
  - Novartis Investigative Site, Incheon
  - Novartis Investigative Site, Seoul
- Spain (14):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Esplugues de Llobregat, Barcelona
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Bilbao, Basque Country
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Alcorcón, Madrid
  - Novartis Investigative Site, Pozuelo de Alarcón, Madrid
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Novartis Investigative Site, Alicante, Valencia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Valencia
- Taiwan (3):
  - Novartis Investigative Site, Taoyuan District, Taiwan
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
- Thailand (3):
  - Novartis Investigative Site, Bangkoknoi, Bangkok
  - Novartis Investigative Site, Bangkok, Phayathai
  - Novartis Investigative Site, Bangkok
- Tunisia (3):
  - Novartis Investigative Site, Sfax, Tunusia
  - Novartis Investigative Site, Sousse
  - Novartis Investigative Site, Tunis
- Turkey (Türkiye) (8):
  - Novartis Investigative Site, Istanbul, Pendik
  - Novartis Investigative Site, Istanbul, TUR
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Aydin
  - Novartis Investigative Site, Denizli
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Okmeydanı
  - Novartis Investigative Site, Samsun
- Novartis Investigative Site, London, United Kingdom
- Vietnam (2):
  - Novartis Investigative Site, Hanoi
  - Novartis Investigative Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: Patient Lay Trial Summary — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1561

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1457 participants who completed preceding studies (CQGE031C2302 (NCT03580369), CQGE031C2303 (NCT03580356), CQGE031C2202 (NCT03437278) or CQGE031C1301 (NCT03907878)) entered the screening period. 515 participants with weekly urticaria activity score (UAS7) <16 during screening entered the OBS1 period (treatment-free period). A total of 1033 participants with UAS7≥ 16 during screening or OBS1 period were assigned to 1 of the 2 treatment arms and entered the treatment period.
Groups:
- Ligelizumab 72 mg LIVI -Ligelizumab 120 mg PFS: Participants received 72 mg of ligelizumab liquid in vial (LIVI), subcutaneously, every 4 weeks for the first 12 weeks. Thereafter, participants received 120 mg of ligelizumab pre-filled syringe (PFS), subcutaneously, every 4 weeks for up to 92 additional weeks (continuous or interrupted if the participant entered the observation period 2)
- Ligelizumab 120 mg LIVI -Ligelizumab 120 mg PFS: Participants received 120 mg of ligelizumab liquid in vial (LIVI), subcutaneously, every 4 weeks for the first 12 weeks. Thereafter, participants received 120 mg of ligelizumab pre-filled syringe (PFS), subcutaneously, every 4 weeks for up to 92 additional weeks (continuous or interrupted if the participant entered the observation period 2)
Period: First Half Treatment Period (52 Weeks)
Arm/Group | Ligelizumab 72 mg LIVI -Ligelizumab 120 mg PFS | Ligelizumab 120 mg LIVI -Ligelizumab 120 mg PFS
Started | 290 | 743
Completed | 140 | 369
Not Completed | 150 | 374
Not completed — Study terminated by sponsor | 134 | 322
Not completed — Subject decision | 11 | 28
Not completed — Lost to Follow-up | 4 | 2
Not completed — Adverse Event | 1 | 11
Not completed — Physician Decision | 0 | 3
Not completed — Protocol deviation | 0 | 3
Not completed — Death | 0 | 2
Not completed — Lack of Efficacy | 0 | 2
Not completed — Pregnancy | 0 | 1
Period: Second Half Treatment Period (52 Weeks)
Arm/Group | Ligelizumab 72 mg LIVI -Ligelizumab 120 mg PFS | Ligelizumab 120 mg LIVI -Ligelizumab 120 mg PFS
Started (Participants with Urticaria Activity Score (UAS7)>6 at Week 52 or who relapsed (UAS7 ≥ 16) during the observation period) | 77 | 206
Completed | 1 | 2
Not Completed | 76 | 204
Not completed — Study terminated by sponsor | 71 | 195
Not completed — Subject decision | 5 | 8
Not completed — Lost to Follow-up | 0 | 1
Period: Observation Period 2 (up to 52 Weeks)
Arm/Group | Ligelizumab 72 mg LIVI -Ligelizumab 120 mg PFS | Ligelizumab 120 mg LIVI -Ligelizumab 120 mg PFS
Started (Participants with UAS7 ≤ 6 at Week 52) | 69 | 201
Completed | 24 | 91
Not Completed | 45 | 110
Not completed — Study terminated by sponsor | 45 | 107
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Subject decision | 0 | 1
Period: Follow-up Period (up to 12 or 52 Weeks)
Arm/Group | Ligelizumab 72 mg LIVI -Ligelizumab 120 mg PFS | Ligelizumab 120 mg LIVI -Ligelizumab 120 mg PFS
Started | 180 | 471
Completed | 157 | 407
Not Completed | 23 | 64
Not completed — Subject decision | 16 | 32
Not completed — Physician Decision | 4 | 16
Not completed — Adverse Event | 1 | 6
Not completed — Lost to Follow-up | 0 | 5
Not completed — New therapy for study indication | 2 | 1
Not completed — Lack of Efficacy | 0 | 2
Not completed — Pregnancy | 0 | 1
Not completed — Protocol deviation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ligelizumab 72 mg LIVI -Ligelizumab 120 mg PFS | Ligelizumab 120 mg LIVI -Ligelizumab 120 mg PFS | Total
Number analyzed (Participants) | 290 | 743 | 1033
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.4 (13.98) | 42.8 (14.40) | 42.7 (14.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 190 | 525 | 715
  Male | 100 | 218 | 318
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 209 | 506 | 715
  Black or African American | 1 | 13 | 14
  Asian | 66 | 199 | 265
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  American Indian or Alaska Native | 11 | 20 | 31
  Multiple | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects From Core Studies (CQGE031C2302 and CQGE031C2303), Receiving the Same Dose Regimen as in the Core Studies, With Well-controlled Disease (UAS7 ≤ 6) at Week 12
Description: The Urticaria Activity Score (UAS) is a composite, diary-recorded score with numeric severity intensity ratings (0=none to 3=intense/severe) for the number of wheals (hives) and the intensity of the pruritus (itch) over the past 12 hours (twice daily). The daily UAS is calculated as the average of the morning and evening scores. The UAS7 is the weekly sum of the daily UAS, which is the composite score of the intensity of pruritus and the number of wheals. UAS7 scores ranged from 0 to 42. A higher UAS7 indicated greater urticaria disease activity.
  A minimum of 4 out of 7 daily scores were needed to calculate the UAS7 values. Otherwise, the weekly score was missing for that week.
  The percentage of subjects transitioning from CQGE031C2302 and CQGE031C2303 and receiving the same dose regimen as in the core studies with UAS7≤ 6 at Week 12 was estimated using multiple imputation method. The 95% confidence interval was derived based on the Wilson score method with continuity correction.
Time Frame: Week 12 of the extension study
Population: Ligelizumab retreatment subpopulation: Participants transitioning from core studies (CQGE031C2302 and CQGE031C2303) who received at least one dose of study treatment and were treated with the same dosage of ligelizumab in the extension study as in the two core studies. Only participants with non-missing UAS7 scores (based on the data after the missing data imputation) for Week 12 were included in this analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ligelizumab 72 mg LIVI -Ligelizumab 120 mg PFS | Ligelizumab 120 mg LIVI -Ligelizumab 120 mg PFS
Number analyzed (Participants) | 290 | 276
Percentage of participants | 53.5 [48.72 to 58.54] | 57.5 [52.71 to 62.57]

2. Secondary Outcome: Percentage of Subjects From Core Studies (CQGE031C2302 and CQGE031C2303), Receiving the Same Dose Regimen as in the Core Studies, With Completely Controlled Disease (UAS7 =0) at Week 12
Description: The Urticaria Activity Score (UAS) is a composite, diary-recorded score with numeric severity intensity ratings (0=none to 3=intense/severe) for the number of wheals (hives) and the intensity of the pruritus (itch) over the past 12 hours (twice daily). The daily UAS is calculated as the average of the morning and evening scores. The UAS7 is the weekly sum of the daily UAS, which is the composite score of the intensity of pruritus and the number of wheals. UAS7 scores ranged from 0 to 42. A higher UAS7 indicated greater urticaria disease activity.
  A minimum of 4 out of 7 daily scores were needed to calculate the UAS7 values. Otherwise, the weekly score was missing for that week.
  The percentage of subjects transitioning from core studies (CQGE031C2302 and CQGE031C2303) and receiving the same dose regimen as in the core studies with UAS7 = 0 at Week 12 was estimated using multiple imputation method.
Time Frame: Week 12 of the extension study
Population: Ligelizumab retreatment subpopulation: Participants transitioning from studies CQGE031C2302 and CQGE031C2303 who received at least one dose of study treatment and were treated with the same dosage of ligelizumab in the extension study as in the two core studies (CQGE031C2302 and CQGE031C2303). Only participants with non-missing UAS7 scores (based on the data after the missing data imputation) for Week 12 were included in this analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ligelizumab 72 mg LIVI -Ligelizumab 120 mg PFS | Ligelizumab 120 mg LIVI -Ligelizumab 120 mg PFS
Number analyzed (Participants) | 290 | 276
Percentage of participants | 37.3 [31.63 to 43.04] | 41.5 [35.61 to 47.36]

3. Secondary Outcome: Change From Extension Study Baseline in the UAS7 at Week 12 in All Subjects From Core Studies (CQGE031C2302 and CQGE031C2303) Receiving the Same Dose Regimen as in the Core Studies
Description: The Urticaria Activity Score (UAS) is a composite, diary-recorded score with numeric severity intensity ratings (0=none to 3=intense/severe) for the number of wheals (hives) and the intensity of the pruritus (itch) over the past 12 hours (twice daily). The daily UAS is calculated as the average of the morning and evening scores. The UAS7 is the weekly sum of the daily UAS, which is the composite score of the intensity of pruritus and the number of wheals. UAS7 scores ranged from 0 to 42. A higher UAS7 indicated greater urticaria disease activity. A negative change score from extension study baseline indicates improvement.
  A minimum of 4 out of 7 daily scores were needed to calculate the UAS7 values. Otherwise, the weekly score was missing for that week.
  The absolute change from extension study baseline in the UAS7 at Week 12 was estimated using multiple imputation method.
Time Frame: Extension study baseline (Week 0), Week 12 of the extension study
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Ligelizumab 72 mg LIVI -Ligelizumab 120 mg PFS | Ligelizumab 120 mg LIVI -Ligelizumab 120 mg PFS
Number analyzed (Participants) | 290 | 276
Score on a scale | -19.83 (13.12) | -20.41 (12.94)

4. Secondary Outcome: Change From Extension Study Baseline in the ISS7 at Week 12 in All Subjects From Core Studies (CQGE031C2302 and CQGE031C2303) Receiving the Same Dose Regimen as in the Core Studies
Description: The Itch Severity Score (ISS) was recorded by the subject twice daily in their eDiary, on a scale of 0 (none) to 3 (intense/severe). A weekly score (ISS7) was derived by adding up the average daily scores of the 7 preceding days. The ISS7 ranged from 0 to 21. A higher ISS7 indicated more severe itching. A negative change score from baseline indicates improvement.
  A minimum of 4 out of 7 daily scores were needed to calculate the ISS7 values. Otherwise, the weekly score was missing for that week.
  The absolute change from extension study baseline in the ISS7 at Week 12 in all subjects from core studies (CQGE031C2302 and CQGE031C2303) receiving the same dose regimen as in the core studies was estimated using multiple imputation method.
Time Frame: Extension study baseline (Week 0), Week 12 of the extension study
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Ligelizumab 72 mg LIVI -Ligelizumab 120 mg PFS | Ligelizumab 120 mg LIVI -Ligelizumab 120 mg PFS
Number analyzed (Participants) | 290 | 276
Score on a scale | -9.12 (6.35) | -9.46 (6.55)

5. Secondary Outcome: Change From Extension Study Baseline in the HSS7 at Week 12 in All Subjects From Core Studies (CQGE031C2302 and CQGE031C2303) Receiving the Same Dose Regimen as in the Core Studies
Description: The Hive Severity Score (HSS) was recorded by the subject twice daily in their eDiary, on a scale of 0 (none) to 3 (> 12 hives/12 hours). A weekly score (HSS7) was derived by adding up the average daily scores of the 7 preceding days. The HSS7 ranged from 0 to 21 A higher HSS7 indicated a greater number of hives. A negative change score from baseline indicates improvement.
  A minimum of 4 out of 7 daily scores were needed to calculate the HSS7 values. Otherwise, the weekly score was missing for that week.
  The absolute change from extension study baseline in the HSS7 at Week 12 in all subjects from core studies (CQGE031C2302 and CQGE031C2303) receiving the same dose regimen as in the core studies was estimated using multiple imputation method.
Time Frame: Extension study baseline (Week 0), Week 12 of the extension study
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Ligelizumab 72 mg LIVI -Ligelizumab 120 mg PFS | Ligelizumab 120 mg LIVI -Ligelizumab 120 mg PFS
Number analyzed (Participants) | 290 | 276
Score on a scale | -10.71 (7.50) | -10.95 (7.11)

6. Secondary Outcome: Cumulative Number of Angioedema-free Weeks (AAS7=0) up to Week 12 in All Subjects From Core Studies (CQGE031C2302 and CQGE031C2303) Receiving the Same Dose Regimen as in the Core Studies
Description: The Weekly angioedema activity score (AAS) is a validated tool to assess occurrence of episodes of angioedema. If the subject reported the occurrence of angioedema ("opening question") with "no", AAS score for this day was 0. If "yes" was the answer to the opening question, the subject continued to answer questions about the duration, severity and impact on daily functioning and appearance of the angioedema. A score between 0 and 3 was assigned to every answer field. The AAS7 was the weekly sum of the daily AAS. AAS7 scores ranged from 0-105. Higher score indicated more severe disease.
  AAS7 in all subjects from core studies (CQGE031C2302 and CQGE031C2303) receiving the same dose regimen as in the core studies was estimated using multiple imputation method. The imputed AAS7 = 0 was used for the cumulative number of weeks that subjects achieved AAS7 = 0 response calculation
Time Frame: From extension study baseline (Week 0) up to Week 12 of the extension study
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Weeks
Arm/Group | Ligelizumab 72 mg LIVI -Ligelizumab 120 mg PFS | Ligelizumab 120 mg LIVI -Ligelizumab 120 mg PFS
Number analyzed (Participants) | 290 | 276
Weeks | 9.30 (0.25) | 9.68 (0.27)

7. Secondary Outcome: Percentage of Subjects From Core Studies (CQGE031C2302 and CQGE031C2303), Receiving the Same Dose Regimen as in the Core Studies, With DLQI = 0-1 at Week 12
Description: The Dermatology Life Quality Index (DLQI) is a 10-item dermatology-specific quality of life (QoL) measure. Subjects rated their dermatology symptoms as well as the impact of their skin condition on various aspects of their lives thinking about the previous 7 days. An overall score was calculated and ranged from 0 to 30. Higher scores indicated worse disease-related QoL. A DLQI score of 0 or 1 indicated that there was no impact of a skin disease on the patient's life.
  The percentage of subjects from core studies (CQGE031C2302 and CQGE031C2303) receiving the same dose regimen as in the core studies with DLQI = 0-1 at Week 12 was estimated using multiple imputation method.
Time Frame: Week 12 of the extension study
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ligelizumab 72 mg LIVI -Ligelizumab 120 mg PFS | Ligelizumab 120 mg LIVI -Ligelizumab 120 mg PFS
Number analyzed (Participants) | 290 | 276
Percentage of participants | 45.6 [39.66 to 51.52] | 55.8 [49.77 to 61.79]

8. Secondary Outcome: Percentage of Subjects With Well-controlled Disease (UAS7 ≤ 6) 12 Weeks After Starting Self-administration
Description: The Urticaria Activity Score (UAS) is a composite, diary-recorded score with numeric severity intensity ratings (0=none to 3=intense/severe) for the number of wheals (hives) and the intensity of the pruritus (itch) over the past 12 hours (twice daily). The daily UAS is calculated as the average of the morning and evening scores. The UAS7 is the weekly sum of the daily UAS, which is the composite score of the intensity of pruritus and the number of wheals. UAS7 scores ranged from 0 to 42. A higher UAS7 indicated greater urticaria disease activity.
  A minimum of 4 out of 7 daily scores were needed to calculate the UAS7 values. Otherwise, the weekly score was missing for that week. Missing data was considered as non-responder in the analysis.
  The percentage of subjects with UAS7≤ 6 at Week 24 (i.e., 12 weeks after starting self-administration) was estimated based on observed data.
Time Frame: Week 24 of the extension study
Population: Self-administration subpopulation: Participants transitioning from preceding studies (CQGE031C2302, CQGE031C2303, CQGE031C2202 and CQGE031C1301) who had at least one injection of study treatment with PFS administered by the participant herself/himself or caregiver either in clinic or outside of clinic
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ligelizumab 72 mg LIVI -Ligelizumab 120 mg PFS | Ligelizumab 120 mg LIVI -Ligelizumab 120 mg PFS
Number analyzed (Participants) | 153 | 383
Percentage of participants | 69.4 [60.86 to 77.07] | 69.5 [64.40 to 74.21]

9. Primary Outcome: Percentage of Subjects From Core Studies (CQGE031C2302 and CQGE031C2303), Receiving the Same Dose Regimen as in Core Studies and Who Achieved UAS7≤ 6 at Week 12 in Core Studies, With Well-controlled Disease (UAS7 ≤ 6) at Week 12 of the Extension Study
Description: The Urticaria Activity Score (UAS) is a composite, diary-recorded score with numeric severity intensity ratings (0=none to 3=intense/severe) for the number of wheals and the intensity of the pruritus over the past 12 hours (twice daily). The daily UAS is calculated as the average of the morning and evening scores. The UAS7 is the weekly sum of the daily UAS, which is the composite score of the intensity of pruritus and the number of wheals. UAS7 scores ranged from 0 to 42. A higher UAS7 indicated greater urticaria disease activity.
  A minimum of 4 out of 7 daily scores were needed to calculate the UAS7 values. Otherwise, the UAS7 was missing for that week. Missing data was considered as non-responder.
  The percentage of subjects transitioning from core studies (CQGE031C2302 and CQGE031C2303) and receiving the same dose regimen as in the core studies who achieved UAS7 ≤ 6 at week 12 in the core studies with UAS7≤ 6 at Week 12 of the extension study was estimated based on observed data.
Time Frame: Week 12 of the extension study
Population: Ligelizumab responder retreatment subpopulation: Participants transitioning from core studies (CQGE031C2302 and CQGE031C2303) who received at least one dose of study treatment, were treated with the same dosage of ligelizumab in the extension study as in the two core studies and achieved UAS7 ≤ 6 at week 12 in the core studies. Only participants with non-missing UAS7 scores based on observed data for Week 12 were included in this analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ligelizumab 72 mg LIVI -Ligelizumab 120 mg PFS | Ligelizumab 120 mg LIVI -Ligelizumab 120 mg PFS
Number analyzed (Participants) | 138 | 144
Percentage of participants | 81.9 [74.73 to 87.92] | 82.6 [75.45 to 88.44]

ADVERSE EVENTS:
Time Frame: Treatment-emergent AEs (TEAEs) were assessed from first dose to 16 weeks post-last dose of each period (below): TRT1A: Within the first 12 weeks of treatment (or up to 16 weeks post-last dose if treatment discontinued), up to 0.5 year. TRT1B: From Week 12 to 52 of treatment (or 16 weeks post-last dose if treatment discontinued), up to 1.1 years. TRT2: From Week 52 to 104 of treatment (or 16 weeks post-last dose if treatment discontinued), up to 1.3 years. Entire study: up to 2.5 years
Description: TEAEs: events started after the first dose within 16 weeks of last dose of study treatment, or pre-existing events that increased in severity within 16 weeks after the last dose. TEAEs counted for each treatment period were those with onset after the start of the treatment period or worsening within that period.
  Safety analyses included participants who received at least one dose of study treatment. Subjects were analyzed according to the treatment they actually received.
Groups:
- TRT1A Ligelizumab 72 mg LIVI-ligelizumab 120 mg PFS: AEs collected during the TRT1A period. During this period, participants received 72 mg of ligelizumab LIVI, subcutaneously, every 4 weeks for the first 12 weeks.
- TRT1A Ligelizumab 120 mg LIVI-ligelizumab 120 mg PFS: AEs collected during the TRT1A period. During this period, participants received 120 mg of ligelizumab LIVI, subcutaneously, every 4 weeks for the first 12 weeks
- TRT1A Total: AEs collected during the TRT1A period.
- TRT1B Ligelizumab 72 mg LIVI - Ligelizumab 120 mg PFS: AEs collected during the TRT1B period. During this period, participants previously treated with ligelizumab 72 mg LIVI received 120 mg of ligelizumab PFS, subcutaneously, every 4 weeks from Week 12 to Week 52.
- TRT1B Ligelizumab 120 mg LIVI - Ligelizumab 120 mg PFS: AEs collected during the TRT1B period. During this period, participants previously treated with ligelizumab 120 mg LIVI received 120 mg of ligelizumab PFS, subcutaneously, every 4 weeks from Week 12 to Week 52.
- TRT1B Total: AEs collected during the TRT1B period.
- TRT2 Ligelizumab 72 mg LIVI - Ligelizumab 120 mg PFS: AEs collected during the TRT2 period. During this period, participants previously treated with ligelizumab 72 mg LIVI received 120 mg of ligelizumab PFS, subcutaneously, every 4 weeks for up to 52 weeks.
- TRT2 Ligelizumab 120 mg LIVI - Ligelizumab 120 mg PFS: AEs collected during the TRT2 period. During this period, participants previously treated with ligelizumab 120 mg LIVI received 120 mg of ligelizumab PFS, subcutaneously, every 4 weeks for up to 52 weeks.
- TRT2 Total: AEs collected during the TRT2 period
- Entire Study Ligelizumab 72 mg LIVI - Ligelizumab 120 mg PFS; Entire Study Ligelizumab 120 mg LIVI - Ligelizumab 120 mg PFS; Entire Study Total: AEs collected from first dose of study treatment to 16 weeks of last dose of study treatment.
Arm/Group | TRT1A Ligelizumab 72 mg LIVI-ligelizumab 120 mg PFS | TRT1A Ligelizumab 120 mg LIVI-ligelizumab 120 mg PFS | TRT1A Total | TRT1B Ligelizumab 72 mg LIVI - Ligelizumab 120 mg PFS | TRT1B Ligelizumab 120 mg LIVI - Ligelizumab 120 mg PFS | TRT1B Total | TRT2 Ligelizumab 72 mg LIVI - Ligelizumab 120 mg PFS | TRT2 Ligelizumab 120 mg LIVI - Ligelizumab 120 mg PFS | TRT2 Total | Entire Study Ligelizumab 72 mg LIVI - Ligelizumab 120 mg PFS | Entire Study Ligelizumab 120 mg LIVI - Ligelizumab 120 mg PFS | Entire Study Total
All-Cause Mortality (participants affected / at risk) | 0/288 | 0/745 | 0/1033 | 0/263 | 3/684 | 3/947 | 0/77 | 0/206 | 0/283 | 0/288 | 3/745 | 3/1033
Serious Adverse Events (participants affected / at risk) | 1/288 | 10/745 | 11/1033 | 5/263 | 32/684 | 37/947 | 2/77 | 3/206 | 5/283 | 8/288 | 44/745 | 52/1033
Other Adverse Events (participants affected / at risk) | 12/288 | 65/745 | 77/1033 | 49/263 | 156/684 | 205/947 | 11/77 | 36/206 | 47/283 | 65/288 | 224/745 | 289/1033
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TRT1A Ligelizumab 72 mg LIVI-ligelizumab 120 mg PFS (N=288) | TRT1A Ligelizumab 120 mg LIVI-ligelizumab 120 mg PFS (N=745) | TRT1A Total (N=1033) | TRT1B Ligelizumab 72 mg LIVI - Ligelizumab 120 mg PFS (N=263) | TRT1B Ligelizumab 120 mg LIVI - Ligelizumab 120 mg PFS (N=684) | TRT1B Total (N=947) | TRT2 Ligelizumab 72 mg LIVI - Ligelizumab 120 mg PFS (N=77) | TRT2 Ligelizumab 120 mg LIVI - Ligelizumab 120 mg PFS (N=206) | TRT2 Total (N=283) | Entire Study Ligelizumab 72 mg LIVI - Ligelizumab 120 mg PFS (N=288) | Entire Study Ligelizumab 120 mg LIVI - Ligelizumab 120 mg PFS (N=745) | Entire Study Total (N=1033)
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Meniere's disease (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Drowning (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Fatigue (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Biliary dilatation (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
COVID-19 (Infections and infestations) | 0 | 2 | 2 | 1 | 7 | 8 | 0 | 2 | 2 | 1 | 11 | 12
Chronic tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 2 | 2
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Oral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Vascular encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Chronic spontaneous urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TRT1A Ligelizumab 72 mg LIVI-ligelizumab 120 mg PFS (N=288) | TRT1A Ligelizumab 120 mg LIVI-ligelizumab 120 mg PFS (N=745) | TRT1A Total (N=1033) | TRT1B Ligelizumab 72 mg LIVI - Ligelizumab 120 mg PFS (N=263) | TRT1B Ligelizumab 120 mg LIVI - Ligelizumab 120 mg PFS (N=684) | TRT1B Total (N=947) | TRT2 Ligelizumab 72 mg LIVI - Ligelizumab 120 mg PFS (N=77) | TRT2 Ligelizumab 120 mg LIVI - Ligelizumab 120 mg PFS (N=206) | TRT2 Total (N=283) | Entire Study Ligelizumab 72 mg LIVI - Ligelizumab 120 mg PFS (N=288) | Entire Study Ligelizumab 120 mg LIVI - Ligelizumab 120 mg PFS (N=745) | Entire Study Total (N=1033)
Pyrexia (General disorders) | 2 | 10 | 12 | 5 | 26 | 31 | 0 | 5 | 5 | 7 | 39 | 46
COVID-19 (Infections and infestations) | 4 | 20 | 24 | 28 | 78 | 106 | 6 | 21 | 27 | 38 | 117 | 155
Nasopharyngitis (Infections and infestations) | 3 | 16 | 19 | 8 | 37 | 45 | 2 | 7 | 9 | 12 | 56 | 68
Headache (Nervous system disorders) | 4 | 26 | 30 | 13 | 43 | 56 | 5 | 6 | 11 | 17 | 64 | 81

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-04-09): https://cdn.clinicaltrials.gov/large-docs/43/NCT04210843/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-27): https://cdn.clinicaltrials.gov/large-docs/43/NCT04210843/SAP_001.pdf